CLINICAL TRIAL: NCT05065125
Title: Clinical Usefulness of Digital Single-operator Cholangioscopy (SpyGlass™) for Post-liver Transplant Anastomotic Stricture
Brief Title: Clinical Usefulness of Digital Single-operator Cholangioscopy(SpyGlass™) for Post-liver Transplant Anastomotic Stricture
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sang Hyub Lee, Professor, Seoul National University Hospital
Other Study IDs: H-2105-134-1219
Record Dates: First submitted 2021-09-22; First posted 2021-10-01 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Liver Transplant; Complications; Biliary Duct Obstruction; Anastomosis, Obstructed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LDLT cohort: Living-donor liver transplatation (LDLT) patients with anastomotic biliary stricture
  Interventions: Device: digital single-operator cholangioscopy

INTERVENTIONS:
Device: digital single-operator cholangioscopy — 1. Duodenoscope passes through esophagus and stomach to the papilla of Vater
  2. SpyScope DS Catheter passes through the duodenoscope and into common bile duct
  3. After direct visualization of anastomosis site stricture, guidewire is passed through SpyScope DS Catheter above the stricture site.

SUMMARY:
Liver transplantation (LT) is an essential treatment for end-stage liver disease. Although clinical outcomes of LT recipients have markedly improved, anastomotic biliary strictures (ABS) are still occurred in 10-40% of post-LT patients.

In the Korea, living donor LT (LDLT) is the more common than deceased donor LT (DDLT). When LDLT is performed, the right lobe graft is usually used, and the right anterior and posterior segmental bile ducts (RASD/RPSD) of the graft are reconstructed by the duct-to-duct anastomosis method to the common hepatic duct of the recipient.

When ABS occurs in LDLT recipients, the stricture site is often very tight and twisted. So, conventional endoscopic procedure is challenging and success rate of ERCP for ABS is still unsatisfactory (about 60%). Furthermore, approach to the RPSD is more intricate than that to RASD because the duct opening is located deeper in a posterior aspect. Therefore, despite being able to benefit the patient, bilateral drainage (both RASD and RPSD) is considered to be more difficult and unilateral drainage of RASD is mainly performed.

In 2015, high-resolution cholangioscopy (SpyGlass™) was introduced. The system enables direct visualization of the bile and pancreatic ducts strictures. The 3rd Generation SpyScope DS II Access & Delivery Catheter introduced in 2018, features increased resolution and adjusted lighting to provide physicians with an even better view of the biliary and pancreatic ducts. To date, only several retrospective studies have evaluated the efficacy of SpyGlass for guidewire placement across the ABS and to the best of our knowledge only one prospective study is ongoing (ClinicalTrials.gov NCT #03205072). In that study ABS in both LDLT and DDLT patients are enrolled. Private communications with the Sponsor of this study, however, have reported that only approximately 10% of the cases are LDLT cases. In addition, there is no reported paper about the usefulness of Spyglass for bilateral drainage and its clinical benefit in post LT ABS.

If successful bilateral drainage is performed by using Spyglass, it may be more helpful for patients than unilateral drainage as it allows sufficient drainage of the transplanted liver. With this prospective study, we intends to investigate the efficacy of Spyglass for bilateral drainage of ABS in LDLT patients and improve drainage success rate. This results can be used as clinical basis for further studies such as randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 or older
* Patients who treated with LDLT (Duct-to-duct anastomosis)
* Patients with confirmed anastomosis site biliary stricture using cross-sectional imaging study (CT, MRI/MRCP).

Exclusion Criteria:

* Patients with age 18 or under
* Pregnant woman
* Patients unable to endoscopic (transpapillary) approach due to prior surgical history
* Patients who did not provide informed consent to participation in the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: LDLT patients with anastomotic biliary stricture
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-10-05 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Rate of Technical success | During endoscopic treatment (ERCP with SpyGlass)
  ① Successful guidewire placement across the stricture site or
  ② Successful subsequent treatment (advancement of dilatation balloon and/or placement of biliary endoprosthesis across the stricture when intended).

SECONDARY OUTCOMES:
Rate of Clinical success | after a month of ERCP procedure
  Rate of improvement of abdominal pain, obstructive jaundice or infection at one month after treatment
Rate of Complication rate | after a month of ERCP procedure
  post-procedural cholangitis, pancreatitis, bleeding, or perforation
Rate of Recurrence rate | after a month of ERCP procedure
  re-intervention within 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Cho IR, Lee SH, Kang J, Kim J, Lee TS, Lee MH, Lee MW, Choi JH, Paik WH, Ryu JK, Kim YT, Hong SK, Choi Y, Yi NJ, Lee KW, Suh KS. Digital single-operator cholangioscopy for difficult anastomotic biliary strictures in living donor liver transplant recipients after failure of standard ERCP: SPYPASS-2 study (with videos). Gastrointest Endosc. 2025 May;101(5):979-987.e3. doi: 10.1016/j.gie.2024.11.017. Epub 2024 Nov 16. PMID 39557203